CLINICAL TRIAL: NCT02088216
Title: Effect of N-acetylcysteine on Exacerbations of Bronchiectasis (BENE): a Randomized Controlled Trial
Brief Title: Effect of Long-term, High-dose N-acetylcysteine on Exacerbations of Bronchiectaisis
Acronym: BENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qian Qi, assistant director, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCFB-FLS-01
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2017-12

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: N-acetylcysteine；; Bronchiectasis；; Acute exacerbations；; Antioxidant；; Anti-inflammatory
MeSH Terms: conditions — Bronchiectasis | interventions — Acetylcysteine

ARMS (2):
- N-Acetylcysteine group (Active Comparator): Participants received 600 mg of oral N-acetylcysteine BID for 12 months.
  Interventions: Drug: N-acetylcysteine
- Control group (Other): Participants received as-needed therapy.
  Interventions: Other: On-demand treatment

INTERVENTIONS:
Drug: N-acetylcysteine — 600mg po twice a day for 12 months
  Arms: N-Acetylcysteine group
Other: On-demand treatment — receive as-needed therapy
  Arms: Control group

SUMMARY:
Objective: To evaluate whether long-term oral N-acetylcysteine as an expectorant drug can reduce the frequency of acute exacerbations of patients with non-cystic fibrosis bronchiectasis and improve their quality of life.

Methods: Patients with non-cystic fibrosis bronchiectasis will be randomly assigned to the observer group (participants receive 600 mg of oral N-acetylcysteine BID for 12 months) or the control group (participants receive oral tablet BID for 12 months). The primary endpoint was the frequency of acute exacerbations.

Expected results: Compared with the control group, the frequency of acute exacerbations of the observer Group will decrease significantly.

Hypothesis: Long-term oral N-acetylcysteine can reduce the frequency of acute exacerbations of patients with non-cystic fibrosis bronchiectasis and improve their quality of life.

DETAILED DESCRIPTION:
Objective: N-acetylcysteine is a classic mucolytic agent. This study aimed to investigate the efficacy and safety of N-acetylcysteine on the risk of exacerbations in bronchiectasis patients.

Methods: A prospective, randomized, controlled trial was conducted between April 1, 2014 and December 31, 2016 in five general hospitals in Shandong Province, China. Adult bronchiectasis patients with at last two exacerbations in the past year were potentially eligible. Patients were randomly assigned to receive oral N-acetylcysteine (600 mg, twice daily, 12 months) or on-demand treatment.

Results: A total of 161 patients were eligible for randomization (81 to the N-acetylcysteine group and 80 to the control group). During the 12-month follow-up, the incidence of exacerbations in the N-acetylcysteine group was significantly lower than that in the control group (1.31 vs. 1.98 exacerbations per patient-year; risk ratio, 0.41; 95% CI, 0.17-0.66; P = 0.0011). The median number of exacerbations in the N-acetylcysteine group was 1 (0.5-2), compared with 2 (1-2) in the control group (U=-2.95, P = 0.003). No severe adverse events were reported in the intervention group.

Conclusion: The long-term use of N-acetylcysteine is able to reduce the risk of exacerbations for bronchiectasis patients.

ELIGIBILITY:
Inclusion Criteria:

1. subjects were aged 18-80 years old;
2. a diagnosis of idiopathic or post-infective bronchiectasis was made;
3. patients had at least two exacerbations in the past year and were in a stable state for at least 4 weeks prior to the primary enrollment.

Exclusion Criteria:

Patients were excluded if they fulfilled any of the following criteria: current smokers; cigarette smoking within 6 months; cystic fibrosis or other etiologies (such as immunodeficiency, allergic bronchopulmonary aspergillosis, traction bronchiectasis caused by emphysema, advanced pulmonary fibrosis, etc.); pulmonary function test results showing a forced expiratory volume in 1 s (FEV1) ≤ 30% of the predicted value; a history of severe cardiovascular or neurological disease; comorbidity with liver disease, kidney disease, malignant tumor, gastric ulcer, or intestinal malabsorption; a known allergy to N-acetylcysteine; pregnancy or lactation (for women); a history of prior macrolide use of more than 1 week; and poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Li, Professor, Study Director — Director
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Qi Q, Ailiyaer Y, Liu R, Zhang Y, Li C, Liu M, Wang X, Jing L, Li Y. Effect of N-acetylcysteine on exacerbations of bronchiectasis (BENE): a randomized controlled trial. Respir Res. 2019 Apr 11;20(1):73. doi: 10.1186/s12931-019-1042-x. PMID 30975143

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine Group: Participants received oral N-acetylcysteine (600 mg, twice daily, 12 months).
- Control Group: Participants received on-demand treatment.
Period: Overall Study
Arm/Group | N-acetylcysteine Group | Control Group
Started | 81 | 80
Completed | 69 | 70
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine Group | Control Group | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.28 (11.90) | 56.56 (12.41) | 54.91 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 52 | 97
  Male | 36 | 28 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Exacerbations
Description: An exacerbation of bronchiectasis is defined as either a change in one or more of the common symptoms of bronchiectasis (sputum volume or purulence, dyspnea, cough, and fatigue/malaise) or the onset of new symptoms (fever, pleurisy, haemoptysis or need for antibiotic treatment).
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: exacerbations
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
exacerbations | 1 [0.5 to 2] | 2 [1 to 2]

2. Secondary Outcome: Change of Volume of Sputum From Baseline Parameters After the 12-month Follow-up.
Description: The change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
mL | -6.46 (22.93) | -18.28 (25.69)

3. Secondary Outcome: Change of Number of Patients With a Positive Sputum Culture for Pseudomonas Aeruginosa
Description: The values in the table were calculated as the value at baseline minus the value at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
Participants | 8 | 5

4. Secondary Outcome: Change of Chronic Obstructive Pulmonary Disease Assessment Test (CAT) Scores From Baselines
Description: Chronic Obstructive Pulmonary Disease Assessment Test (CAT) scores: the minimum value is 0 and the maximum value is 40.
  0-10 points: "slight impact"; 11-20 points: "medium impact"; 21-30 points: "serious impact"; 31-40 points: "very serious impact".
  The change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
score on a scale | -3.79 (5.40) | -1.44 (6.19)

5. Secondary Outcome: Change in Percentage of Predicted Forced Expiratory Volume in One Second (FEV1%) From Baselines
Description: as for outcome 2
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
percentage of predicted FEV1 | 1.16 (16.50) | 0.13 (7.78)

6. Secondary Outcome: Change of Forced Expiratory Volume in One Second (FEV1) (L) From Baselines
Description: as for outcome 2
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: L
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
L | -0.10 (0.37) | 0.03 (0.16)

7. Secondary Outcome: Change of Forced Vital Capacity (FVC) From Baselines
Description: as for outcome 2
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: L
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
L | 0.01 (0.46) | 0.03 (0.22)

8. Secondary Outcome: Time to the First Exacerbation
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
days | 140 [95.90 to 184.10] | 115 [77.75 to 152.25]

9. Secondary Outcome: Time to Recurrent Exacerbations
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
days | 313.70 [297.05 to 330.36] | 266.88 [244.60 to 289.15]

10. Secondary Outcome: Nature of Sputum (Number of Patients With Yellow Purulent)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
Participants | 12 | 31

11. Secondary Outcome: Adverse Events (AEs) (Elevation of Liver Enzymes)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine Group | Control Group
Number analyzed (Participants) | 81 | 80
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | N-acetylcysteine Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/81 | 3/80
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 8/81 | 6/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine Group (N=81) | Control Group (N=80)
Epigastric discomfort (Gastrointestinal disorders) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02088216/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02088216/SAP_001.pdf